CLINICAL TRIAL: NCT03575806
Title: A Single-center, Open-label, Exploratory Trial of Autologous Immunotherapy for Hepatocellular Carcinoma (HCC) With Microvascular Invasion (MVI) After Radical Resection
Brief Title: Combine TACE and Autologous Tcm Immunotherapy Versus TACE Alone for HCC With MVI After Radical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hong Zhao, assistant director physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CancerIHCAMS-HCC-Tcm
Record Dates: First submitted 2018-06-12; First posted 2018-07-03 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma; Malignant Neoplasm
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE+Tcm group (Experimental): Experimental arm: TACE plus autologous Tcm immunotherapy to treat HCC.
  Interventions: Combination Product: TACE plus autologous Tcm immunotherapy
- TACE group (Active Comparator): Active comparator: TACE to treat HCC.
  Interventions: Procedure: TACE

INTERVENTIONS:
Combination Product: TACE plus autologous Tcm immunotherapy — TACE:transcatheter arterial chemoembolization.
  Autologous Tcm immunotherapy: to collect patient's own immune cells and then given back to the patient after amplified in vitro.
  Arms: TACE+Tcm group
Procedure: TACE — TACE:transcatheter arterial chemoembolization.
  Arms: TACE group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of combining autologous Tcm immunotherapy and TACE in HCC patients with MVI after radical resection. Patients will be assigned either to the experimental arm to receive autologous Tcm immunotherapy and TACE or to the active comparator (TACE alone).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the common cancer worldwide, which is the third cause of cancer related deaths. Radical hepatic resection remains the main treatment for hepatocellular carcinoma, the 5-year survival rate of HCC after surgery was 60-70%. Unfortunately, HCC is prone to postoperative recurrence that more than 50% of patients relapse within 2 years, which has become the key to restrict the therapeutic effect of hepatocellular carcinoma. Microvascular invasion (MVI) is one of the main risk factors for poor prognosis in HCC.

Autologous cell immunotherapy is to collect patient's own immune cells and then given back to the patient after amplified in vitro that can improve the anti-tumor immune response. Tcm (central memory T cells) are effective anti-tumor immune cells that exhibit the long-term survival and self-renewal capacity in vivo. Autologous Tcm immunotherapy combining chemotherapy, surgery or radiotherapy would effectively prolong survival period, prevent tumor recurrence and metastasis, then improve quality of life in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study.
2. Subject has accepted radical hepatic resection, and preoperative imaging is no vascular invasion.
3. Postoperative pathology confirmed Hepatocellular carcinoma with negative margin and microvascular invasion (MVI).
4. Age between 18-75 years old.
5. Radiology confirmed complete response (CR) after radical surgery.
6. Child-Pugh A.
7. Eastern Cooperative Oncology Group(ECOG) body condition score 0.
8. Adequate hepatic and renal function:

   Hemoglobin ≥ 9.0g/dl. Absolute neutrophil count (ANC) > 1,500/mm3. Platelets ≥ 50,000/ul. Total bilirubin (TBIL) ≤ 2mg/dl. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 the upper limit of normal (ULN) for the institution.

   Alkaline phosphatase (ALP) ≤ 4 the upper limit of ULN. Prothrombin time (PT) > 50% or prothrombin time-international normalized ratio (PT-INR) < 2.3.

   Serum creatinine (CREA) ≤ 1.5 the upper limit of ULN.
9. Female subjects have had a negative blood pregnancy test within 2 week,
10. Subjects be willing to use appropriate contraception during the trial and 2 weeks after the last administration of immunotherapy.
11. Radiology such as CT and MRI were performed in 4 weeks before the study.

Exclusion Criteria:

1. Recurrent HCC.
2. Portal vein embolus.
3. Cardiovascular disease:

   Evidence of NYHA functional class III or IV heart disease. Unstable coronary artery disease (CAD) is not allowed, while Myocardial Infarction (MI) 6 months of starting study is allowed.

   Cardiac arrhythmias requiring antiarrhythmic drugs except β-blockers or digoxin are not allowed.

   Uncontrolled hypertension.
4. History of Human Immunodeficiency Virus (HIV) or syphilis infection.
5. Severe inflammation, NCI CTCAE Version 3.0 grade > 2.
6. Epilepsy requiring steroid or antiepileptic drugs.
7. History of allotransplantation.
8. History or any evidence of hemorrhage.
9. Subjects undergoing renal dialysis.
10. Pregnancy or breast-feeding.
11. Prior or undergoing cancers that primary sites are different from the carcinoma of this study. Exceptions to this are:

    Cervical carcinoma in situ (CIS) Cured basal cell carcinoma Superficial bladder tumor Cured cancers over 3 years before the study
12. Uncontrolled Ascites by diuretic treatment.
13. History of encephalopathy.
14. Gastrointestinal hemorrhage in 30 days before the study.
15. History of esophageal variceal hemorrhage and it is no effective treatment to prevent the recurrence of hemorrhage.
16. Major surgery except radical hepatic resection was performed in 4 weeks before the study.
17. Autologous bone marrow transplantation (ABMT) in 4 weeks before the study.
18. Concurrent treatment on another clinical trial or treatment on another clinical trial in 4 weeks before the study.
19. Drug abuse, medical treatment, mental illness or social disorders that would interfere with subjects' participation, or confound the results of the trial.
20. Any condition that would interfere with or endanger the safety and compliance of subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhao, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai J, Zhao J, Liu D, Xie H, Qi H, Ma J, Sun Z, Zhao H. Efficacy and Safety of Central Memory T Cells Combined With Adjuvant Therapy to Prevent Recurrence of Hepatocellular Carcinoma With Microvascular Invasion: A Pilot Study. Front Oncol. 2021 Dec 3;11:781029. doi: 10.3389/fonc.2021.781029. eCollection 2021. PMID 34926296

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was not of a randomized design, patients were recruited by their willingness to receive the Tcm transfusion as the adjuvant therapy after screening and meeting the eligibility criteria. As pathological classification with MVI was determined after 1 week postoperatively, patients consented with radical operation would be screened again.
Groups:
- TACE Group: Control arm: only TACE
  (TACE: transcatheter arterial chemoembolization)
- TACE+Tcm Group: Experimental arm: TACE plus autologous Tcm immunotherapy
  (TACE:transcatheter arterial chemoembolization)
  Autologous Tcm immunotherapy: collected patient's own immune cells and then transfused back to patient after being amplified in vitro.
Period: Overall Study
Arm/Group | TACE Group | TACE+Tcm Group
Started | 25 | 27
Completed | 25 | 23
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Per Protocol Set (PPS):
  1. Be eligiable for inclusion criterial and exclusion criterial;
  2. Complete the whole follow-up program;
  3. Refuse other therapies for HCC in the follow-up program which would influence the efficacy evaluation of Tcm.
Groups:
- Total: Total of all reporting groups
Arm/Group | TACE Group | TACE+Tcm Group | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 17 | 41
  >=65 years | 1 | 6 | 7
Age, Continuous [Mean (Full Range); unit: years] | 53.4 [27 to 68] | 53.7 [31 to 77] | 53.5 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 19 | 16 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 25 | 23 | 48
Eastern Cooperative Oncology Group(ECOG) [Count of Participants; unit: Participants] — ECOG STATUS
  0, Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  Participants
    ECOG=0 | 25 | 23 | 48
    ECOG=1 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS) Time
Description: Recurrence-free survival was defined as the interval (in months) between hepatectomy and diagnosis of recurrence using either intrahepatic recurrence or extrahepatic metastasis.
Time Frame: 12 months
Population: PPS (Per Protocol Set)
Measure: Median (Standard Deviation); unit: months
Arm/Group | TACE Group | TACE+Tcm Group
Number analyzed (Participants) | 25 | 23
months | 9.5 (3.99) | 12 (3.24)

2. Secondary Outcome: Overall Survival (OS) Rate at 24 Months
Description: Overall survival rate = the number of patients in TACE/TACE+Tcm group survived at 24 months/the number of total patients assigned into TACE/TACE+Tcm group.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TACE Group | TACE+Tcm Group
Number analyzed (Participants) | 25 | 23
Participants
  Survival | 25 | 23
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: Laboratory examination of blood tests, liver and kidney function of all patients were collected every 4 weeks during Tcm treatment and every 12 weeks after Tcm treatment in 48 weeks or ended the last follow-up. 1 patients assigned into TACE+Tcm group requested withdrawing without any administration of Tcm.
Groups:
- TACE Group: Control arm: only TACE
  (TACE: TACE:transcatheter arterial chemoembolization)
Arm/Group | TACE Group | TACE+Tcm Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 19/25 | 9/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TACE Group (N=25) | TACE+Tcm Group (N=26)
Hepatic pain (Hepatobiliary disorders) | 19 | 9 — Patients with total bilirubin or ALT or AST elevation
Bone marrow hypocellular (Blood and lymphatic system disorders) | 9 | 0 — patients with decreasing white blood cells or lymphocytes

LIMITATIONS AND CAVEATS:
This study was a pilot study with small sample size, which would influence the statistical results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT03575806/Prot_SAP_ICF_000.pdf